CLINICAL TRIAL: NCT02684721
Title: Does an 8-week Home-based Exercise Programme Affect Physical Capacity, Quality of Life, Sick Leave and Use of Psychoactive Drugs in Patients With Pulmonary Embolism. A Randomised Clinical Trial
Brief Title: Does a Home-based Exercise Programme Affect Physical Capacity and Quality of Life in Patients With Pulmonary Embolism?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Aalborg University Hospital (Other); Horsens Hospital (Other); Regional Hospital West Jutland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6300001
Record Dates: First submitted 2016-01-20; First posted 2016-02-18 (Estimated); Last update posted 2019-08-19 (Actual); Status verified 2016-11

CONDITIONS: Pulmonary Embolism
Keywords: rehabilitation; physical capacity; quality of life
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Patients in the control group receive usual care as a minimum. This includes 3-5 days of hospitalisation where the anticoagulant treatment is initiated. The patient and the relatives receive general information about the disease and the course of treatment, the medication and future prevention of embolism. In the year following discharge the patient is booked for a check-up of their anticoagulant treatment with a physician or a nurse as required.
- Exercise group (Experimental): 8-week home-base exercise programme: Patients in the intervention group receive the same usual care as patients in the control group. In addition the patients participate in an 8 week home-based exercise programme, including follow-up telephone calls with the physiotherapist after 1 week, 2 weeks and 4 weeks. Briefly put, the patients are required to exercise for a minimum of 3 times per week for 30-60 minutes, and with 3-4 intervals of approximately 1 minute at a high intensity level. Total exercise time and intervals increase during the 8 week programme. The patients can choose whatever type of exercise they prefer, and they are generally encouraged to choose something they already do, or something that they have previously had positive experiences doing.
  Interventions: Other: 8-week home-based exercise programme

INTERVENTIONS:
Other: 8-week home-based exercise programme — 8-week home-based exercise programme is assigned to patients in exercise group following discharge. This includes 3 follow-up telephone calls by physiotherapist.
  Arms: Exercise group

SUMMARY:
In a randomised design the study aims to investigate whether an intervention of 8 weeks home-based exercise in addition to usual care can positively influence the physical capacity, quality of life, sick leave and use of psychoactive drugs in patients medically treated for pulmonary embolism.

DETAILED DESCRIPTION:
Background: The existing knowledge regarding pulmonary embolism is primarily focused on the diagnostic methods and medical treatment of the condition, and furthermore on the short term prognosis in terms of mortality and complications. Very few studies investigate how every day life is affected in patients struck by a pulmonary embolism, although many patients display worries and concerns about their physical, emotional and social well-being after discharge. For the time being, no rehabilitation options are available for these patients in Denmark.

Methods and materials: 140 patients medically treated for pulmonary embolism will be recruited from 6 different hospitals. After inclusion the patients will be randomly allocated to either the control group, receiving usual care, or the intervention group, receiving an 8-week home-based exercise programme in addition to usual care. At the time of inclusion, after 2 months and after 6 months, the patients' physical capacity is measured using the Incremental Shuttle Walk test.

Furthermore the patients' complete a questionnaire on quality of life (EQ-5D and Pulmonary Embolism Quality of Life Questionnaire), self-reported sick leave and use of psychoactive drugs. All follow-up measurements and visits take place at the hospital from which the patient was discharged.

Expected outcome and perspective: The investigators expect that the home-based exercise programme will improve the overall treatment outcome for the patients in the intervention group. The study will furthermore contribute significantly to the limited knowledge about the optimal rehabilitation for this group of patients, and may thereby form the basis of future recommendations in this field.

ELIGIBILITY:
Inclusion Criteria:

* Objectively verified acute pulmonary embolism
* Treatment with anticoagulant drugs
* 18-70 years of age
* Competency in the Danish language

Exclusion Criteria:

* Pulmonary embolism as a secondary finding in relation to scan performed due to another disease.
* Severe co-morbidity (malignant, inflammatory or psychiatric)
* Unable to perform the Incremental Shuttle Walk test for other reasons (e.g. amputation or intermittent claudication).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Incremental Shuttle Walk test from baseline to 6 months after baseline | Baseline, 2 months and 6 months after baseline
  Validated outcome measure for assessing a person's maximum walking capacity

SECONDARY OUTCOMES:
Change in Pulmonary Embolism Quality of Life from baseline to 6 months | Baseline, 2 months and 6 months after baseline
  Disease specific quality of life questionnaire, developed for patients with pulmonary embolism. Validated in a Scandinavian setting.
Change in EuroQol 5 Dimensions (EQ-5D) from baseline to 6 months | Baseline, 2 months and 6 months after baseline
  Generic quality of life questionnaire. Validated in Danish, including Danish preference values
Sick leave in the past 4 weeks measured at 2 and 6 month follow-up | Baseline, 2 months and 6 months after baseline
  The patients are required to state the number of days on sick leave within the last 4 weeks, according to the following categories: No days off work, less than 5 days off work, less than 10 days off work, 10 days or more off work.
Average weekly use of psychoactive drugs in the past 4 weeks measured at 2 and 6 month follow-up | Baseline, 2 months and 6 months after baseline
  The patients are required to state their average weekly use of psychoactive drugs within the last 4 weeks according to the following categories: No days per week, 1-4 days per week, 5-7 days per week.

CONTACTS AND LOCATIONS:
Overall Officials: Nanna Rolving, PhD, Principal Investigator — Diagnostic Centre, Regional Hospital Silkeborg, Silkeborg, Denmark
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Regional hospital Herning, Herning
  - Diagnostic Centre, Regional Hospital Silkeborg, Silkeborg

REFERENCES:
- [Background] Rolving N, Brocki BC, Mikkelsen HR, Ravn P, Bloch-Nielsen JR, Frost L. Does an 8-week home-based exercise program affect physical capacity, quality of life, sick leave, and use of psychotropic drugs in patients with pulmonary embolism? Study protocol for a multicenter randomized clinical trial. Trials. 2017 May 30;18(1):245. doi: 10.1186/s13063-017-1939-y. PMID 28558825
- [Background] Rolving N, Brocki BC, Andreasen J. Coping with everyday life and physical activity in the aftermath of an acute pulmonary embolism: A qualitative study exploring patients' perceptions and coping strategies. Thromb Res. 2019 Oct;182:185-191. doi: 10.1016/j.thromres.2019.06.007. Epub 2019 Jun 19. PMID 31262439
- [Derived] Rolving N, Brocki BC, Bloch-Nielsen JR, Larsen TB, Jensen FL, Mikkelsen HR, Ravn P, Frost L. Effect of a Physiotherapist-Guided Home-Based Exercise Intervention on Physical Capacity and Patient-Reported Outcomes Among Patients With Acute Pulmonary Embolism: A Randomized Clinical Trial. JAMA Netw Open. 2020 Feb 5;3(2):e200064. doi: 10.1001/jamanetworkopen.2020.0064. PMID 32108888